CLINICAL TRIAL: NCT05784311
Title: Standard Versus Pre-emptive Antibiotic Treatment to Reduce the Rate of Infectious Outcomes After Whipple's Procedure (SPARROW): a Multicenter, Randomized Controlled Trial
Brief Title: Standard Versus Prolonged Antibiotic Prophylaxis After Pancreatoduodenectomy (SPARROW)
Acronym: SPARROW
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Leiden University Medical Center (Other)
Responsible Party: Principal Investigator, J.S.D. Mieog, MD PhD, Principal Investigator, Leiden University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL82304.058.22
Record Dates: First submitted 2023-02-27; First posted 2023-03-24 (Actual); Last update posted 2024-10-21 (Actual); Status verified 2024-10

CONDITIONS: Pancreatic Cancer
Keywords: Antibiotic prophylaxis; Preoperative biliary drainage; Surgical site infection
MeSH Terms: conditions — Pancreatic Neoplasms; Surgical Wound Infection | interventions — Cefuroxime; Metronidazole

STUDY DESIGN:
Intervention Model Description: Patients will be randomized with a 1:1 allocation before surgery into the intervention or control group:
  * Patients in the intervention group will receive perioperative prophylaxis (similar to the control group) followed by five days of 1500mg IV cefuroxime and 500mg IV metronidazole thrice daily.
  * Patients in the control group will only receive perioperative prophylaxis (a single dose of 5-7mg/kg gentamicin followed by 2gr IV cefazolin and 500mg IV metronidazole every 4h of surgery), which will be discontinued after surgery.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Perioperative plus prolonged antibiotic prophylaxis (Experimental): Prolonged prophylaxis: a single dose of 5-7mg/kg gentamicin followed by 2gr IV cefazolin and 500mg IV metronidazole every 4 hours of surgery (perioperative prophylaxis) followed by five days of 1500mg IV cefuroxime and 500mg IV metronidazole thrice daily
  Interventions: Drug: Cefuroxime; Drug: Metronidazole
- Only perioperative prophylaxis (No Intervention): Perioperative prophylaxis: a single dose of 5-7mg/kg gentamicin followed by 2gr IV cefazolin and 500mg IV metronidazole every 4 hours of surgery.

INTERVENTIONS:
Drug: Cefuroxime — 1500mg IV cefuroxime thrice daily during five days.
  Other Names: Zinacef
  Arms: Perioperative plus prolonged antibiotic prophylaxis
Drug: Metronidazole — 500mg IV metronidazole thrice daily during five days.
  Other Names: Flagyl
  Arms: Perioperative plus prolonged antibiotic prophylaxis

SUMMARY:
The goal of this multicenter randomized controlled trial is to evaluate the additional value of pre-emptive antibiotic treatment on clinically relevant organ/space surgical site infections (OSIs) in patients undergoing pancreatoduodenectomy with a high risk for contaminated bile. The main objectives it aims to answer are:

* To evaluate the effect of pre-emptive antibiotic prophylaxis on clinically relevant OSIs in patients undergoing pancreatoduodenectomy with a high risk for contaminated bile
* To evaluate the effect of pre-emptive antibiotic prophylaxis on other postoperative outcomes (e.g. OSIs, superficial SSIs, POPF, PPH, major morbidity, ICU admission, readmission, length of hospital stay, and mortality).
* To evaluate concordance between perioperatively obtained bile cultures and postoperative cultures from infectious sites, and to evaluate antibiotic sensitivity patterns of the cultured microorganisms.

Participants will be randomized with a 1:1 allocation before surgery into the intervention or control group:

* Patients in the intervention group will receive perioperative prophylaxis (similar to the control group) followed by five days of 1500mg IV cefuroxime and 500mg IV metronidazole thrice daily.
* Patients in the control group will only receive perioperative prophylaxis (a single dose of 5-7mg/kg gentamicin followed by 2gr IV cefazolin and 500mg IV metronidazole every 4h of surgery), which will be discontinued after surgery.

DETAILED DESCRIPTION:
Rationale: The additional value of pre-emptive antibiotic treatment after pancreatoduodenectomy is undetermined as previous research reported conflicting results regarding infectious complications. Prolonged antibiotic prophylaxis (formally pre-emptive antibiotic treatment) after pancreatoduodenectomy might reduce the rate of surgical site infections in patients with a high risk for contaminated bile (predominantly patients with preoperative biliary drainage or an ampullary malignancy). Current national and international guidelines lack clear recommendations regarding pre-emptive antibiotic treatment leading to substantially varying antibiotic prophylactic regimes between institutes.

Objective: This trial evaluates the additional value of pre-emptive antibiotic treatment on clinically relevant organ/space surgical site infections (OSIs) in patients undergoing pancreatoduodenectomy with a high risk for contaminated bile.

Study design: This multicenter, randomized controlled, superiority trial compares perioperative versus pre-emptive antibiotic treatment during five postoperative days after pancreatoduodenectomy in patients with a high risk for contaminated bile.

Study population: Adult patients undergoing pancreatoduodenectomy with a high risk for contaminated bile (patients with preoperative biliary drainage or an ampullary malignancy). Patients with a contraindication for the study antibiotics or a preoperative indication for antibiotics (e.g. cholangitis of preoperative abscesses) are excluded.

Intervention: Participants will be randomized to either perioperative prophylaxis (cefazolin, metronidazole and a single dose of 5-7mg/kg gentamicin, control arm) or additional cefuroxime and metronidazole for five postoperative days (experimental arm).

Main study endpoints: The primary endpoint are organ/space infections (OSIs) within 90 days after surgery requiring a therapeutic intervention. Secondary endpoints are OSIs, isolated OSIs, wound infections, postoperative pancreatic fistula, bile or enteric anastomotic leakage, post pancreatectomy hemorrhage, delayed gastric emptying, bacteremia, Clostridium difficile infection, major morbidity (Clavien-Dindo ≥III), reintervention, ICU admission, length of hospital stay, readmission, and in-hospital and 90-day mortality. Besides, switch of postoperative antibiotics, antibiotic sensitivity patterns and concordance between perioperative bile and postoperative surgical site cultures are analyzed.

Sample size: The sample size is calculated for superiority to achieve an OSI difference of 15% (40% vs 25%). With a 80% power (1-β) and a two-sided significance level (α) of 5.0%, a sample of 304 evaluable patients is required for superiority. Assuming a 3% non-resection rate due to metastatic disease and a 3% loss-of-follow-up rate, an expected number of 322 included patients are needed to reach the sample size of 304 evaluable patients to demonstrate superiority for the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective pancreatoduodenectomy with a high risk for contaminated bile defined as patients with preoperative biliary drainage or an ampullary malignancy.
* Age >18 years

Exclusion Criteria:

* Pregnancy
* Contraindication for the study antibiotics (e.g. allergy or intolerance)
* Preoperative planned therapeutic antibiotic treatment (i.e. for cholangitis or liver abscesses)
* A reduced renal function, defined as an eGFR of <60 ml/min/1.73m2 measured on the closest timepoint prior to pancreatoduodenectomy

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 344 (Estimated)
Dates: Start 2023-03-06 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Rate of clinically relevant organ/space surgical site infection (OSI) between patients with perioperative versus prolonged antibiotic prophylaxis | 90 days after surgery
  A clinically relevant OSI is defined by the following criteria:
  * A deep surgical site infection involving any part of the abdomen (e.g. organs and/or spaces) other than the surgical incision within 90 days after surgery.
  * AND Requires radiological, endoscopic or surgical intervention OR therapeutic antibiotics required for an episode of sepsis, defined as two or more SIRS criteria.
  * AND Organisms isolated from an aseptically obtained culture.

SECONDARY OUTCOMES:
The rate of organ/Space Infection (OSI) between patients with perioperative versus prolonged antibiotic prophylaxis | 90 days
  An OSI is defined by the CDC definition:
  o The infection appears to be related to the operative procedure and infection involves any part of the anatomy (e.g., organs or spaces) other than the incision opened or manipulated during the operative procedure, and at least one of the following is present:
  1. Purulent drainage from a drain that is placed into the organ/space.
  2. Organisms isolated from an aseptically obtained culture of fluid or tissue in the organ/space.
  3. An abscess or other evidence of infection involving the organ/space on direct examination, during reoperation, or by histopathologic or radiologic examination.
  4. Diagnosis of an organ/space SSI by a surgeon or attending physician."
The rate of isolated OSI between patients with perioperative versus prolonged antibiotic prophylaxis | 90 days
  Isolated OSI is defined as an OSI without concurrent anastomotic leakage (pancreatojejunostomy, hepaticojejunostomy or gastrojejunostomy). The concept of an isolated OSI is used to separately classify abdominal infections without concurrent anastomotic leakage.
The rate of superficial incisional SSI between patients with perioperative versus prolonged antibiotic prophylaxis | 90 days
  A superficial surgical site infection after surgery which involves superficial or deep soft tissue (skin, muscle or fascia, but no intra-abdominal tissue), and at least one of the following criteria is present:
  * Purulent drainage from the incision or subcutaneous tissue.
  * Isolation of microorganisms from an aseptically obtained culture of fluid or tissue from the superficial incision of subcutaneous tissue.
  * Superficial infections of the skin or subcutaneous tissue which is deliberately opened by a surgeon or attending physician OR at least one of the following signs are present: localizes pain, tenderness, swelling, heat or fever >38 degrees).
The rate of clinically relevant postoperative pancreatic fistula between patients with perioperative versus prolonged antibiotic prophylaxis | 90 days
  Grade B or C postoperative pancreatic fistula (POPF) defined by the International Study Group of Pancreatic Surgery definition:
  Grade A: Amylase >3 times upper limit of the institutional normal serum amylase value
  Grade B: Grade A + persistant drainage >3 weeks, clinically relevant change in management of POPF, percutaneous or endoscopic drainage, angiographic procedures for bleeding, or signs of infection without organ failure.
  Grade C: Grade A or B requiring reoperation, resulting in organ failure or death.
The rate of bile leakage between patients with perioperative versus prolonged antibiotic prophylaxis | 90 days
  Grade A, B or C defined by the ISGLS definition:
  Grade A: Bile leakage requiring no or little change in patients' clinical management.
  Grade B: Bile leakage requiring a change in patients clinical management (eg, additional diagnostic or interventional procedures) but manageable without relaparotomy, or a Grade A bile leakage lasting for >1 week.
  Grade C: Bile leakage requiring relaparotomy
The rate of post pancreatectomy hemorrhage between patients with perioperative versus prolonged antibiotic prophylaxis | 90 days
  Grade A, B or C defined by the ISGPS definition:
  Grade A: Early (<24h after surgery), intra- or extraluminal, clinically mild.
  Grade B: Early (<24h after surgery), intra- or extraluminal and clinically severe OR later (>24h after surgery), intra- or extraluminal and clincally mild.
  Grade C: Late (>24h after surgery), intra- or extraluminal and clinically severe.
The rate of delayed gastric emptying between patients with perioperative versus prolonged antibiotic prophylaxis | 90 days
  Grade A, B or C defined by the ISGPS definition:
  Grade A: Until day 4-7 or replacement of feeding tube > 3 days after surgery
  Grade B: Until day 8-14 or replacement of feeding tube > 7 days after surgery
  Grade C: >day 14 or replacement of feeding tube > 14 after surgery
The rate of postoperative bacteremia between patients with perioperative versus prolonged antibiotic prophylaxis | 90 days
  Defined as a positive blood culture obtained during a septic period (defined as two or more SIRS criteria)
The rate of Clostridium difficile infection between patients with perioperative versus prolonged antibiotic prophylaxis | 90 days
  Defined by a positive fecal culture for Clostridium difficile
Rate of major complications between patients with perioperative versus prolonged antibiotic prophylaxis | 90 days
  Major complications is defined by a Clavien-Dindo score of ≥III.
  Clavien-Dindo classification of Surgical Complications:
  Grade I: Any deviation from the normal postoperative course without the need for pharmacological treatment or surgical, endoscopic and radiological interventions.
  Grade II: Requiring pharmacological treatment with drugs other than such allowed for grade I complications.
  Grade IIIa: Requiring surgical, endoscopic or radiological intervention not under general anesthesia Grade IIIb: Requiring surgical, endoscopic or radiological intervention under general anesthesia
  Grade IVa: Life-threatening complication (including CNS complications)* requiring IC/ICU-management with single organ dysfunction (including dialysis).
  Grade IVb: Life-threatening complication (including CNS complications)* requiring IC/ICU-management with multi organ dysfunction.
  Grade V: Death of a patient
The number of reinterventions in patients with perioperative versus prolonged antibiotic prophylaxis | 90 days
  Reinterventions could be either radiological, surgical or endoscopic reinterventions
The number of ICU admission in patients with perioperative versus prolonged antibiotic prophylaxis | 90 days
  ICU admission
Length of hospital stay in patients with perioperative versus prolonged antibiotic prophylaxis | 90 days
  In days
The number of readmissions between patients with perioperative versus prolonged antibiotic prophylaxis | 90 days
  Readmission into the hospital
Mortality | 90 days
  In-hospital and 90-days mortality

OTHER OUTCOMES:
The percentage of patients with a deviation from antibiotic study protocol | 5 days
  Study protocol:
  * Control arm: Perioperative antibiotic prophylaxis (cefazolin, metronidazole and single-dose gentamicin).
  * Intervention arm: Perioperative plus prolonged antibiotics (cefuroxime and metronidazole for five postoperative days).
Antibiotic sensitivity patterns of microorganisms cultured from bile cultures and postoperative cultures from infectious sites between patients with perioperative versus prolonged antibiotic prophylaxis | 90 days
  Rate of Antibiotic sensitivity patterns in bile cultures and cultures from surgical sites
The percentage of concordance of microorganisms in bile and cultures from infectious sites postoperatively | 90 days
  Defined as the similarity of microorganisms between perioperative bile cultures and postoperative cultures from infectious sites.

CONTACTS AND LOCATIONS:
Overall Officials: J. Sven D. Mieog, MD PhD, Principal Investigator — Leiden University Medical Center
Locations (11):
- Netherlands (11):
  - Leiden University Medical Center, Leiden, South Holland
  - Jeroen Bosch Ziekenhuis, 's-Hertogenbosch
  - Amsterdam University Medical Center, Amsterdam
  - Amphia Ziekenhuis, Breda
  - Catharina Ziekenhuis, Eindhoven
  - Medisch Spectrum Twente, Enschede
  - Groningen University Medical Center, Groningen
  - Maastricht University Medical Center, Maastricht
  - Radboud University Medical Center, Nijmegen
  - Erasmus MC Cancer Institute, Rotterdam
  - Regional Academic Cancer Center Utrecht, Utrecht

IPD SHARING:
Plan to Share IPD: No
Available upon request to the principal investigator